CLINICAL TRIAL: NCT02517567
Title: Pilot Study on the Effect of Daily Disposable Silicone Hydrogel Contact Lenses on Tear Film Lipids
Brief Title: DAILIES TOTAL1® - Comparative Assessment of Tear Film Evaporation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLT978-P001
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Results first posted 2018-02-01 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-07

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sequence 1 (Other): Delefilcon A, then narafilcon A, then somofilcon A, then no lens wear. Each contact lens product was worn for 8 hours. The 'No Lens wear' treatment was evaluated over an 8 hour period.
  Interventions: Device: Delefilcon A contact lenses; Device: Narafilcon A contact lenses; Device: Somofilcon A contact lenses
- Sequence 2 (Other): Narafilcon A, then no lens wear, then delefilcon A, then somofilcon A. Each contact lens product was worn for 8 hours. The 'No Lens wear' treatment was evaluated over an 8 hour period.
  Interventions: Device: Delefilcon A contact lenses; Device: Narafilcon A contact lenses; Device: Somofilcon A contact lenses
- Sequence 3 (Other): Somofilcon A, then delefilcon A, then no lens wear, then narafilcon A. Each contact lens product was worn for 8 hours. The 'No Lens wear' treatment was evaluated over an 8 hour period.
  Interventions: Device: Delefilcon A contact lenses; Device: Narafilcon A contact lenses; Device: Somofilcon A contact lenses
- Sequence 4 (Other): No lens wear, then somofilcon A, then narafilcon A, then delefilcon A. Each contact lens product was worn for 8 hours. The 'No Lens wear' treatment was evaluated over an 8 hour period.
  Interventions: Device: Delefilcon A contact lenses; Device: Narafilcon A contact lenses; Device: Somofilcon A contact lenses

INTERVENTIONS:
Device: Delefilcon A contact lenses — Daily disposable, silicone hydrogel contact lenses used according to manufacturer's instructions
  Other Names: DAILIES TOTAL1®
Device: Narafilcon A contact lenses — Daily disposable, silicone hydrogel contact lenses used according to manufacturer's instructions
  Other Names: 1-DAY ACUVUE® TruEye®
Device: Somofilcon A contact lenses — Daily disposable, silicone hydrogel contact lenses used according to manufacturer's instructions
  Other Names: clariti® 1 day

SUMMARY:
The purpose of this study is to evaluate the tear film evaporation of symptomatic soft contact lens wearers in the absence of contact lens wear and after at least 8 hours of contact lens wear.

DETAILED DESCRIPTION:
This study consists of 5 visits (1 screening, 4 assessment) with a maximum of 6 days between assessment visits and at least 24 hours of no lens wear the day prior to the visit. Each subject will be randomized to a crossover sequence of 4 periods. Different study lenses will be worn during 3 of the periods, for at least 8 hours each, and the remaining period will have no lens wear.

ELIGIBILITY:
Inclusion Criteria:

* Sign an informed consent document;
* Adapted, current soft contact lens wearer;
* Symptoms of contact lens discomfort as defined by the Symptomatology (Eligibility) Questionnaire;
* Can be successfully fitted with study lenses;
* Willing to wear lenses for a minimum of 8 hours prior to each study visit;
* Willing to discontinue artificial tears and rewetting drops usage on the days of study visits;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear;
* Use of systemic or ocular medications for which contact lens wear could be contraindicated as determined by the investigator;
* Monocular (only 1 eye with functional vision) or fit with only one lens;
* History of herpetic keratitis, ocular surgery, or irregular cornea;
* Known pregnancy and lactation;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2016-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, Clinical Trial Management, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 study center located in Australia.
Pre-assignment Details: Of the 37 enrolled, 7 subjects were exited as screen failures prior to randomization and 1 subject discontinued after randomization prior to exposure to the investigational product. This reporting group includes all randomized and exposed subjects (29).
Groups:
- Sequence 1: DAILIES TOTAL1 (DT1)/TruEye/clariti/No Lens
- Sequence 2: TruEye/No Lens/DT1/clariti
- Sequence 3: clariti/DT1/No Lens/TruEye
- Sequence 4: No Lens/clariti/TruEye/DT1
Period: First Exposure (8 Hours)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 8 | 7 | 8
Completed | 6 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Second Exposure (8 Hours)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 8 | 7 | 8
Completed | 6 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Third Exposure (8 Hours)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 8 | 7 | 8
Completed | 6 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Exposure (8 Hours)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 8 | 6 (One subject discontinued between Period 3 and Period 4 (withdrawal by subject)) | 8
Completed | 6 | 8 | 6 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects/eyes exposed to any investigational product (including the 'No Lens wear' treatment) evaluated in this study, except for lenses used at Visit 1 for the purpose of parameter optimization and fitting, as they were not intended for the assessment of safety and effectiveness (Safety Analysis Set).
Groups:
- Overall: Delefilcon A, narafilcon A, and somofilcon A contact lenses worn bilaterally (in both eyes) and a period of no lens wear in a randomized crossover fashion
Arm/Group | Overall
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (5.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Tear Film Evaporation Rate
Description: Tear film evaporation rate (amount of tears (grams or g) that evaporates over a surface area (m2) per hour (h)) assessment was performed using the VapoMeter as a non-invasive measurement of tear film evaporation over 10 seconds. Measurements were taken on both the right and left eyes after 8 hours of lens wear or no lens wear, as applicable. A higher evaporation rate can be a contributing factor to eye irritation and lens intolerance.
Time Frame: Day 1, Hour 8, each product
Population: This analysis population includes all randomized subjects (Intent-to-Treat). To address the primary objective of comparing Lens vs. No Lens, results from all 3 study lenses are combined. Therefore, subjects (eyes) are counted multiple times in Lens group due to crossover design and number of eyes with non-missing response is reported.
Measure: Mean (Standard Deviation); unit: gm^-2 h
Units Other Than Participants: Eyes
Groups:
- Lens: Delefilcon A contact lenses, narafilcon A contact lenses, and somofilcon A contact lenses worn bilaterally in cross-over fashion as randomized. Each product worn for one day, 8 hours minimum.
- No Lens: One 8-hour day of no lens wear as part of the crossover sequence
Arm/Group | Lens | No Lens
Number analyzed (Participants) | 29 | 29
Number analyzed (Eyes) | 172 | 58
gm^-2 h | 120.88 (45.563) | 105.63 (53.361)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 5 weeks). AEs are reported as pretreatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to exposure to the investigational product (including the 'No Lens wear' treatment)
- DAILIES TOTAL1: All subjects exposed to DT1 contact lenses worn for 8 hours during Period 1, 2, 3, or 4 as randomized
- TruEye: All subjects exposed to TruEye contact lenses worn for 8 hours during Period 1, 2, 3, or 4 as randomized
- Clariti: All subjects exposed to clariti contact lenses worn for 8 hours during Period 1, 2, 3, or 4 as randomized
- No Lens: All subjects exposed to "No lens wear" for 8 hours during Period 1, 2, 3, or 4 as randomized
Arm/Group | Pretreatment | DAILIES TOTAL1 | TruEye | Clariti | No Lens
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/29 | 0/28 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/29 | 0/28 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/37 | 0/29 | 0/28 | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.